CLINICAL TRIAL: NCT04797624
Title: Does Coronavirus Disease 2019 (COVID-19) Pandemic Cause a Delay in the Diagnosis of Gastric Cancer Patients?
Status: Completed | Type: Observational
Sponsor: Adana City Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Şeker, Ahmet Seker, Associate Professor, MD, Department of Gastroenterological Surgery, Adana City Training and Research Hospital
Other Study IDs: 1248
Record Dates: First submitted 2021-03-12; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Stomach Cancer; Corona Virus Infection
Keywords: gastric surgery; COVID-19; SARS-COV-2; pandemic; stomach surgery; cancer surgery
MeSH Terms: conditions — Stomach Neoplasms; Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Baseline group: The baseline group included the patients diagnosed with gastric cancer between January 1, 2019, and December 31, 2019, in the pandemic group at the Adana City Training and Research Hospital, Department of General Surgery, Divisions of Gastroenterological Surgery and Surgical Oncology. Gastric cancer surgery for adequate patients.
  Interventions: Procedure: Gastric cancer surgery
- Pandemic group: The pandemic group included the patients diagnosed with gastric cancer during the period between March 1, 2020, and December 31, 2020, in the pandemic group at the Adana City Training and Research Hospital, Department of General Surgery, Divisions of Gastroenterological Surgery and Surgical Oncology. Gastric cancer surgery for adequate patients.
  Interventions: Procedure: Gastric cancer surgery

INTERVENTIONS:
Procedure: Gastric cancer surgery — Appropriate gastric cancer surgery types for the convenient patients

SUMMARY:
The aim of this study is to analyze whether COVID-19 causes a delay in the diagnosis of gastric cancer patients particularly in the TNM staging of the tumor, or not and to compare the number of newly diagnosed patients with gastric cancer before and during the COVID-19 pandemic period.

DETAILED DESCRIPTION:
The study included the patients diagnosed with gastric cancer during the period between March 1, 2020, and December 31, 2020, in the pandemic group at the Adana City Training and Research Hospital, Department of General Surgery, Divisions of Gastroenterological Surgery and Surgical Oncology. For the baseline group, patients diagnosed with gastric cancer between January 1, 2019, and December 31, 2019, was included in the same department.

Clinical and pathological data of the patients were retrospectively collected from the hospital medical records. The following parameters were compared between the pandemic and baseline periods; age and gender distributions, mean monthly numbers of newly diagnosed patients, CEA and CEA-19.9 levels, the type of the surgery, the location of the tumor, the frequency of the patients receiving neoadjuvant treatment, American Society of Anesthesiologists (ASA) score, length of the hospital stay, clinical staging and pathologic TNM staging.

ELIGIBILITY:
Inclusion Criteria:

Patients newly diagnosed with gastric cancer at specified intervals will be included in the study.

Exclusion Criteria:

* Having an additional second primary tumor

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: newly diagnosed gastric cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Comparison of the mean monthly numbers of newly diagnosed gastric cancer patients between the groups | from March 1, 2020 to December 31, 2020 -from January 1, 2019 to December 31, 2019
  numbers of newly diagnosed gastric cancer
Comparison of the clinical staging and pathologic TNM staging of the patients | from March 1, 2020 to December 31, 2020 -from January 1, 2019 to December 31, 2019
  Clinical staging was determined based on the results of a physical exam, biopsy, and imaging tests including computed tomography (CT), PET CT, endoscopy and the endoscopic ultrasound. Surgical stage refers to the pathologic stage of the surgical specimen determined based on the American Joint Committee on Cancer (AJCC) TNM system.

SECONDARY OUTCOMES:
Comparison of the demographic data | from March 1, 2020 to December 31, 2020 -from January 1, 2019 to December 31, 2019
  age and gender distributions, mean monthly numbers of newly diagnosed patients, CEA and CEA-19.9 levels, the type of the surgery, the location of the tumor, the frequency of the patients receiving neoadjuvant treatment, American Society of Anesthesiologists (ASA) score, length of the hospital stay,

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Seker, MD, Principal Investigator — Adana City Training and Research Hospital
Locations (1):
- Adana City Training and Research Hospital, Adana, Yuregir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feletto E, Grogan P, Nickson C, Smith M, Canfell K. How has COVID-19 impacted cancer screening? Adaptation of services and the future outlook in Australia. Public Health Res Pract. 2020 Dec 9;30(4):3042026. doi: 10.17061/phrp3042026. PMID 33294902
- [Background] Vecchione L, Stintzing S, Pentheroudakis G, Douillard JY, Lordick F. ESMO management and treatment adapted recommendations in the COVID-19 era: colorectal cancer. ESMO Open. 2020 May;5(Suppl 3):e000826. doi: 10.1136/esmoopen-2020-000826. PMID 32457036
- [Background] Dinmohamed AG, Visser O, Verhoeven RHA, Louwman MWJ, van Nederveen FH, Willems SM, Merkx MAW, Lemmens VEPP, Nagtegaal ID, Siesling S. Fewer cancer diagnoses during the COVID-19 epidemic in the Netherlands. Lancet Oncol. 2020 Jun;21(6):750-751. doi: 10.1016/S1470-2045(20)30265-5. Epub 2020 Apr 30. No abstract available. PMID 32359403